CLINICAL TRIAL: NCT07288333
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Efficacy, Safety, Tolerability, and Pharmacokinetics of NBI-1117570 in Adults With Schizophrenia Who Warrant Inpatient Hospitalization
Brief Title: Evaluation of NBI-1117570 in Inpatient Adults With Schizophrenia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NBI-1117570-SCZ2035; 2025-521868-35-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; NBI-1117570
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- NBI-1117570: Lower-dose (Experimental): Participants will receive a lower-dose of NBI-1117570.
  Interventions: Drug: NBI-1117570
- NBI-1117570: Higher-dose (Experimental): Participants will receive a higher-dose of NBI-1117570.
  Interventions: Drug: NBI-1117570
- Placebo (Placebo Comparator): Participants will receive placebo matched to NBI-1117570.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NBI-1117570 — Oral administration
  Arms: NBI-1117570: Higher-dose; NBI-1117570: Lower-dose
Drug: Placebo — Oral administration
  Arms: Placebo

SUMMARY:
The primary objective for this study is to evaluate the efficacy of NBI-1117570 compared with placebo on improving behavioral and psychological symptoms of schizophrenia in adults who warrant inpatient hospitalization.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 55 years of age
* Primary diagnosis of schizophrenia ≥1 year before screening.
* Participant is experiencing an acute exacerbation or relapse of symptoms with onset less than 2 months before screening and currently requires hospitalization.
* Participant must have had a positive response to at least 1 antipsychotic therapy (other than clozapine) for the treatment of a prior acute relapse.

Key Exclusion Criteria:

* Considered to be at imminent risk of suicide or injury to self or others.
* History of epilepsy, seizures, or convulsions.
* Has orthostatic hypotension, or history of pulmonary hypertension, obstructive coronary artery disease, hypertrophic cardiomyopathy, myocardial infarction, coronary artery revascularization, heart failure, left ventricular hypertrophy, moderate or severe cardiac valvopathy, or other cardiovascular conditions or measures that would preclude participation.
* Currently taking prohibited medications.
* Pregnant or lactating.

Note: Additional inclusion/exclusion criteria may apply, per protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Day 35 | Day 35

SECONDARY OUTCOMES:
Number of Participants With Treatment-emergent Adverse Event (TEAEs) | Day 1 up to Day 49

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences

IPD SHARING:
Plan to Share IPD: No